CLINICAL TRIAL: NCT01131052
Title: Diabetes Care in Nursing Home Residents: A Randomized Controlled Study
Brief Title: Diabetes in the Elderly: Prospective Study
Acronym: DMElderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guillermo Umpierrez (Other)
Responsible Party: Sponsor-Investigator, Guillermo Umpierrez, Professor of Medicine, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00038789
Record Dates: First submitted 2010-05-19; First posted 2010-05-26 (Estimated); Results first posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes; Hyperglycemia
Keywords: elderly populations; diabetes
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia | interventions — Insulin Glargine; Insulin; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BASAL PLUS (Active Comparator): Diabetic subjects receive insulin glargine once daily plus corrective doses of insulin glulisine before meals and bedtime as needed
  Interventions: Drug: Insulin Glargine; Drug: Insulin glulisine
- sliding scale regular insulin (SSRI) (Active Comparator): Diabetic subjects receive sliding scale regular insulin (SSRI) before meals and at bedtime as needed
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin Glargine — glargine once a day
  Other Names: Lantus
  Arms: BASAL PLUS
Drug: Insulin — sliding scale regular insulin (SSRI) given before meals and at bedtime as needed
  Other Names: Novolin R
  Arms: sliding scale regular insulin (SSRI)
Drug: Insulin glulisine — glulisine given as needed before meals
  Other Names: Apridra
  Arms: BASAL PLUS

SUMMARY:
Diabetes is highly prevalent in the elderly, afflicting about 20% of older adults aged 65-75 years and 40% of adults >80years of age. It is expected that the number of elderly people suffering from diabetes will increase in the future, as general life expectancy is increasing.

Nursing home residents with diabetes have higher rates of serious comorbidities and have greater activity of daily living dependencies than other residents without diabetes. In addition, persons with diabetes have higher risk of hypertension, heart disease, stroke depression, cognitive impairment, and cardiovascular mortality than individuals without diabetes.

There are a few retrospective studies in elderly patients analyzing quality of diabetes care and glycemic control adjusted for medications and presence of co-morbidities in long-term care facilities; however, no previous randomized controlled trials have demonstrated benefits of glycemic control on clinical outcome, quality of life, and rate of acute metabolic complications (hyperglycemia and hypoglycemic events) in long-term care facilities. In addition, it is not known whether the use of basal insulin is superior to treatment with sliding scale insulin (SSI) in long-term care facility residents with type 2 diabetes.

Accordingly, the investigators propose to conduct a prospective randomized control trial comparing the efficacy and safety of the basal (glargine) insulin regimen and sliding scale regular insulin in the management of nursing home patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females > 60 years of age.
2. Blood glucose > 150 mg/dl and A1C > 7.5%.
3. A known history of T2DM, receiving either diet alone, oral monotherapy, or with any combination of oral antidiabetic agents (metformin, sulfonylureas, repaglinide, nateglinide, pioglitazone, rosiglitazone, sitagliptin).
4. Patients admitted for non-cardiac elective or emergency surgery or trauma.

Exclusion Criteria:

1. Subjects with increased blood glucose concentration, but without a known history of diabetes (stress hyperglycemia).
2. Subjects with a history of diabetic ketoacidosis and hyperosmolar hyperglycemic state (26).
3. Patients with clinically relevant hepatic disease (diagnosed liver cirrhosis and portal hypertension), corticosteroid therapy, or impaired renal function (creatinine ≥ 3.5 mg/dl).
4. Patients with recognized or suspected endocrine disorders associated with increased insulin resistance, acromegaly, or hyperthyroidism

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory SOM
Locations (1):
- Guillermo Umpierrez, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Pasquel FJ, Powell W, Peng L, Johnson TM, Sadeghi-Yarandi S, Newton C, Smiley D, Toyoshima MT, Aram P, Umpierrez GE. A randomized controlled trial comparing treatment with oral agents and basal insulin in elderly patients with type 2 diabetes in long-term care facilities. BMJ Open Diabetes Res Care. 2015 Aug 28;3(1):e000104. doi: 10.1136/bmjdrc-2015-000104. eCollection 2015. PMID 26336609

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at Emory University-Wesley Woods Campus between March 2011 through December 2013.
Groups:
- BASAL PLUS: Diabetic subjects receive glargine once daily plus corrective doses of glulisine before meals and bedtime as needed
Period: Overall Study
Arm/Group | BASAL PLUS | Sliding Scale Regular Insulin (SSRI)
Started | 75 | 75
Completed | 75 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BASAL PLUS | Sliding Scale Regular Insulin (SSRI) | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 73 | 72 | 145
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 47 | 96
  Male | 26 | 28 | 54
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With a Mean Blood Glucose Concentration of Less Than 70 mg/dL
Description: Mean weekly blood glucose concentration less than 70 mg/dL at 3 months
Time Frame: 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Basal Plus | Sliding Scale Regular Insulin (SSRI)
Number analyzed (Participants) | 75 | 75
percentage of participants | 28 | 31

2. Primary Outcome: Percent of Participants With a Mean Blood Glucose Concentration of Less Than 40 mg/dL
Description: Mean weekly blood glucose concentration less than 40 mg/dL at 3 months
Time Frame: 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Basal Plus | Sliding Scale Regular Insulin (SSRI)
Number analyzed (Participants) | 75 | 75
percentage of participants | 0 | 1

3. Secondary Outcome: Mean Blood Glucose Concentration
Description: Mean blood glucose concentration at baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Basal Plus | Sliding Scale Regular Insulin (SSRI)
Number analyzed (Participants) | 75 | 75
mg/dL | 198.2 (39.7) | 191.8 (35.2)

4. Secondary Outcome: Mean of Glycosylated Hemoglobin (hbA1c)
Description: Mean glycosylated hemoglobin (hbA1c) at baseline. The A1C test result is reported as a percentage. The higher the percentage, the higher a person's blood glucose levels have been. A normal A1C level is below 5.7 percent.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percent of glycosylated hemoglobin
Arm/Group | Basal Plus | Sliding Scale Regular Insulin (SSRI)
Number analyzed (Participants) | 75 | 75
percent of glycosylated hemoglobin | 6.8 (0.8) | 6.5 (0.7)

5. Secondary Outcome: Mean of Daily Blood Glucose Concentration
Description: Mean of daily blood glucose concentration at baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Basal Plus | Sliding Scale Regular Insulin (SSRI)
Number analyzed (Participants) | 75 | 75
mg/dL | 163.0 (29.4) | 137.7 (27.4)

6. Secondary Outcome: Mean of Glycosylated Hemoglobin (hbA1c)
Description: as for outcome 4
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percent of glycosylated hemoglobin
Arm/Group | Basal Plus | Sliding Scale Regular Insulin (SSRI)
Number analyzed (Participants) | 75 | 75
percent of glycosylated hemoglobin | 7.0 (1) | 6.3 (1.0)

7. Secondary Outcome: Mean of Glycosylated Hemoglobin (hbA1c)
Description: as for outcome 4
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percent of glycosylated hemoglobin
Arm/Group | Basal Plus | Sliding Scale Regular Insulin (SSRI)
Number analyzed (Participants) | 75 | 75
percent of glycosylated hemoglobin | 6.7 (1.1) | 6.3 (0.7)

8. Primary Outcome: Mean of Weekly Fasting Blood Glucose Concentration
Description: Mean weekly blood glucose concentration at 3 months
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Basal Plus | Sliding Scale Regular Insulin (SSRI)
Number analyzed (Participants) | 75 | 75
mg/dL | 130 (26) | 123 (23)

ADVERSE EVENTS:
Arm/Group | BASAL PLUS | Sliding Scale Regular Insulin (SSRI)
Serious Adverse Events (participants affected / at risk) | 9/75 | 12/75
Other Adverse Events (participants affected / at risk) | 17/75 | 23/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BASAL PLUS (N=75) | Sliding Scale Regular Insulin (SSRI) (N=75)
Death (Cardiac disorders) | 1 | 0 — Severe Aortic Stenosis
ER visit (Cardiac disorders) | 2 | 1
Hospitalization (Cardiac disorders) | 6 | 11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BASAL PLUS (N=75) | Sliding Scale Regular Insulin (SSRI) (N=75)
Infection (Infections and infestations) | 11 | 16
ARF (Renal and urinary disorders) | 2 | 6
CV (Cardiac disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes